CLINICAL TRIAL: NCT05005832
Title: Influence of Walking Pilgrimage on Changes in Body Composition, Biochemical Parameters, Circulatory and Respiratory Efficiency and Foot Biomechanics in Healthy Women and Men of All Ages.
Status: Completed | Type: Observational
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Szczepan Wiecha, Principal Investigator, Józef Piłsudski University of Physical Education
Other Study IDs: SKE 01-25/2021
Record Dates: First submitted 2021-07-23; First posted 2021-08-16 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Cardiovascular Diseases; Health Behavior; Foot Injuries and Disorders; Skin Condition
MeSH Terms: conditions — Cardiovascular Diseases; Health Behavior; Foot Injuries; Disease; Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People participating in the walking pilgrimage: People taking part in the study will be healthy people without any existing systemic diseases and musculoskeletal injuries, and will not engage in professional physical activity. The age of the respondents will be in the range of 18-65 years and BMI in the range of 18-39. People who have valid medical examinations will be admitted to the tests, with no contraindications to physical activity.
  Interventions: Other: multi day walking

INTERVENTIONS:
Other: multi day walking — Over the course of 14 days, the pilgrims will cover a distance of about 300 km.

SUMMARY:
The aim of the study is to assess the health habits and changes in body composition and exercise capacity as well as blood biochemical parameters of people participating in 14-21-day walking pilgrimages. This type of physical activity can be classified as long-term and multi-stage hiking tours. Among the people participating in the pilgrimage, a significant part of the population are people aged> 50 years. Moderate physical activity is an important pro-health element, however, it has not been determined yet how long and accumulated activity may affect the health of pilgrims. Suddenly taking up activity and the challenge of walking several hundred kilometres may be a heavy burden for the body, and its effects may have a negative impact on the body. The evaluation of the processes taking place in the body under the influence of this type of physical activity, motivated by religious goals, will expand the scope of knowledge about safety as well as health indications and contraindications for this type of activity. It will also allow identifying adaptive changes and their effects

ELIGIBILITY:
Inclusion Criteria:

women and men aged 18-65

BMI (body mass index) at the level of 18-39

Exclusion Criteria:

Chronic diseases Musculoskeletal injuries Mental disorders Surgery or hospitalization in the last year before the start of the study Pregnancy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People taking part in a walking pilgrimage from Biała Podlaska to Częstochowa (Poland) over a distance of approximately 350 kilometres and a duration of approximately 14 days in August 2021
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Systematic Coronary Risk Evaluation | 14-21 days
  Systematic Coronary Risk Evaluation scales (SCORE) are high and low cardiovascular risk charts based on gender, age, total cholesterol, systolic blood pressure and smoking status, with relative risk chart, qualifiers and instructions.
  SCORE calculate 10-year risk of fatal cardiovascular disease (%),
  * Low- to moderate-risk persons (calculated SCORE <5%)
  * High-risk persons (calculated SCORE >5% and <10%):
  * Very-high-risk persons (calculated SCORE >10%):
  Charts are available free at https://www.escardio.org/Education/Practice-Tools/CVD-prevention-toolbox/SCORE-Risk-Charts
  Risk estimation using SCORE: https://www.heartscore.org/en_GB/access-heartscore-quick-calculator

SECONDARY OUTCOMES:
Tiffeneau-Pinelli index | 14-21 days
  Tiffeneau-Pinelli index FEV1/FVC% The FEV1/FVC ratio, also called Tiffeneau-Pinelli index, is a calculated ratio represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).The result of this ratio is expressed as FEV1%.
  Normal FEV1% values are approximately 70-80%
Clarke angle | 14-21 days
  The Clarke angle (CL)enables the assessment of the longitudinal arch of the foot. Feet having a CL angle value of less than 42° are classified as the feet with the fallen arch, i.e., the flatfoot (pes planus), feet classified as having a proper (normal) arch are characterised by the CL restricted within the range of 42-54° (pes rectus), whereas feet having CL ≥ 55° are classified as feet with a high arch (pes cavus)
Transepidermal water loss | 14-21 days
  Transepidermal water loss (TEWL) is the most widely used objective measurement for assessing the barrier function of skin in healthy individuals. TEWL is the quantity of condensed water that diffuses across a fixed area of stratum corneum to the skin surface per unit time.
  TEWL are stated as grams of water per square meter per hour (g/m2/h). Measured at forehead and right cheek.
  TEWL normal values (mean,95% CI) for forehead 12.8 (11.7-14.0) and cheek 13.9 (12.9-14.9).

CONTACTS AND LOCATIONS:
Locations (1):
- Jozef Pilsudski University of Physical Education in Warsaw Faculty in Biala Podlaska, Biała Podlaska, Poland